CLINICAL TRIAL: NCT02986334
Title: Brain Mechanisms For Clinical Placebo in Chronic Pain: A Randomized Clinical Trial of Placebo, Active Treatment, and No Treatment in Chronic Back Pain
Brief Title: Placebo In Chronic Back Pain (Phase 2)
Acronym: PICP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Apkar Apkarian (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Apkar Apkarian, Professor in Physiology, Anesthesiology and Physical Medicine and Rehabilitation, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00080585 (Phase 2); 5R01AT007987-03 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Chronic Low Back Pain
Keywords: chronic; low back; back; pain; brain; MRI
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Pain | interventions — Naproxen; Omeprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Treatment Intervention (No Intervention): Observational Subjects randomized to this arm will be asked to discontinue their current pain medications for the length of the study. This arm is not blinded, as both study staff and participants will be aware that they are not receiving a study treatment.
- Active Treatment Intervention (Active Comparator): Naproxen & Omeprazole Subjects randomized to this arm will be asked to discontinue their current pain medications and take one 500mg naproxen capsule and one 40mg omeprazole capsule twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants is receiving (blind to active versus placebo treatment).
  Interventions: Drug: Naproxen; Drug: Omeprazole
- Placebo Treatment Intervention (Placebo Comparator): Subjects randomized to this arm will be asked to discontinue their current pain medications and take two placebo capsules twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants is receiving (blind to active versus placebo treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Subjects enrolled in the active treatment arm will receive 500mg of Naproxen prescribed twice daily, once in the morning and evening.
  Other Names: Aleve; Anaprox; Antalgin; Feminax Ultra; Flanax; Inza; Midol Extended Relief; Nalgesin; Naposin; Naprelan; Naprogesic; Naprosyn; Narocin; Proxen; Soproxen; Synflex; Xenobid
  Arms: Active Treatment Intervention
Drug: Omeprazole — Subjects enrolled in the active treatment arm will receive 20mg of Omeprazole prescribed twice daily, once in the morning and evening. Furthermore, subjects should take this one hour before a meal.
  Other Names: Prilosec; Iosepine
  Arms: Active Treatment Intervention
Drug: Placebo — Subjects enrolled in the inactive treatment arm will receive two prescriptions, however, there are no active ingredients and are intended to look identical to the active treatment. Therefore, subjects will be instructed exactly the same way as if they were ingesting the active treatment.
  Other Names: Sugar Pill
  Arms: Placebo Treatment Intervention

SUMMARY:
This study is designed to examine brain properties for placebo response in chronic back pain patients. The investigators have preliminary data indicating that, in blinded clinical trial studies with neutral instructions regarding treatment, chronic back pain (CBP) patients can be subdivided into placebo responders and non-responders, and these differences are PREDICTABLE a priori, by brain activity. The results imply that CBP placebo may have clinical utility and that its properties can be studied by human brain imaging techniques. In Phase I of the study, the investigators seek to identify brain imaging parameters that predict the propensity for the placebo response in an independent CBP cohort. In Phase II, the investigators will evaluate the interaction between placebo response and medication treatment in individuals stratified as placebo responders versus non-responders. This research is designed to critically assess the neurobiology of placebo analgesia for chronic pain in a partially-blind clinical trial.

DETAILED DESCRIPTION:
Visit 1 (week -3): Screening visit (90 min):

Participants will be evaluated with inclusion/exclusion criteria and complete the informed consent documents. A medical/pain history will be taken and physical exam will be completed by a physician and participants will be asked to rate their current back pain intensity. Participants will complete a set of 10 questionnaires that will ask about health and medical history, past and current pain levels, personality, and emotions. Participants will be allowed to take breaks and walk around during this time so that participants don't get tired while filling out questionnaires. Finally, participants will have blood drawn for screening purposes including to see if kidneys and liver are functioning as they should (the investigators will take 40 mL or about 8 teaspoons). Participants will be asked to return in 2 weeks for baseline magnetic resonance imaging (MRI) scans. Participants will be asked to discontinue current pain medications 14 days prior to Visit 2 and take only the rescue medication ("rescue" medication that is also known as acetaminophen/Tylenol ®), given for pain during this time (see below) - this is so that the investigators can assess baseline amount of pain. Participants will be informed that they may be randomized in the placebo group and/or the no-treatment group (Visit 3) once one qualifies to continue in the study. Participants must, therefore,a be willing and able to stop taking the medication for pain for up to a maximum of 12 weeks during this study. Participants will be given acetaminophen (500 mg, up to 4 times per day) to take for pain relief (as rescue medication), a dose that can be continued throughout the study. Participants are free to stop participation at any point in the study. Participants randomized into the treatment arm may receive the anti-inflammatory drug naproxen, since it is known to increase the risk of stomach and intestinal side effects, a combined naproxen/esomeprazole drug regimen will be given to participants to provide some protection for these types of side effects.

Visit 2 (week -1): Baseline Scan (90 min):

Participants will rate their pain intensity, complete questionnaires, and undergo brain scanning (anatomical and functional scans). Participants will receive medication, which can be used if the pain becomes too much to handle (500 mg four times per day maximum). The researcher will ask participants about how often participants used the "rescue" medication and any changes in health they may have experienced since the last visit.

Visit 3 (week 0): Start of Treatment Period and Randomization (30-45 min):

Participants will rate their pain intensity and complete questionnaires. Participants will be randomized into either a drug (placebo or naproxen and esomeprazole) treatment group or no treatment group; if participants are assigned to a treatment group (active or placebo), neither participants nor the clinical coordinator/assistant will know which group participants are allocated in. Enough medication will be given to participants to last until the next visit. The placebo group will receive two placebo capsules twice daily and the active drug group will receive one naproxen capsule (500mg) and one esomeprazole capsule (20mg) twice daily (morning and night) for the treatment period. The medication (Naproxen or Placebo) needs to be taken with at least one full glass (8 oz) of water and the other medication (Esomeprazole or Placebo) should be taken one hour before a meal. The researcher will provide the study medication; if participants were randomized into the no treatment group, participants will only receive rescue medication. The researcher will ask participants about how often participants used the "rescue" medication and any side effects participants experienced since Visit 2 took place. Additional "rescue" medication will be given.

Visit 4 (week 3): Continuing Assessment (30-45 min). The procedures described for Visit 3 will be repeated during this visit. The researcher will ask participants about how often they used the "rescue" medication and any side effects experienced since Visit 3 took place. As well, the researcher will ask how often participants took the study medication (if in a treatment group) and document the total pills ingested.

Visit 5 (week 6): End of Treatment/Start of Washout and Final Scan (60-90 min):

The procedures described for Visit 2 will be repeated during this visit. The researcher will ask participants about how often and reliably participants took the medication (if in a treatment group), as well as how often they used the "rescue" medication and any side effects experienced since Visit 4 took place. Participants will only receive the "rescue" medication for the upcoming 3 weeks.

Visit 6 (week 9): Final Visit/End of Washout (30-45 min):

Participants will return to complete questionnaires, but no brain scans will be done. The researcher will ask participants about how often they used the "rescue" medication and any side effects experienced since Visit 5 took place. If participants are in one of the treatment groups, participants will be asked to return all of the study medication and rescue medication at this time, and all treatment will be stopped at this visit.

ELIGIBILITY:
Inclusion Criteria:

* History of low back pain for a minimum of 6 months with or without signs and symptoms of radiculopathy
* Male or female, between the ages of 18 and 75 years, with no racial or ethnic restrictions
* Must have a Visual Analog Scale (VAS) pain score of 5 mm (of 10 mm maximum) at the screening visit (for which 0mm = no pain, and 10 mm = worst pain imaginable);
* Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires;
* Must be in generally stable health;
* Must sign an informed consent document after a complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate
* Must have, on average, 5/10 units (VAS scale) of pain over the course of a two-week period prior to visit 1; rounding up from 4.5/10 is permissible.
* Must be willing to complete daily smart phone/computer app ratings.

Exclusion Criteria:

* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills;
* Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, fibromyalgia, history of tumor in the back;
* Other comorbid chronic pain or neurological conditions;
* Involvement in litigation regarding their back pain or having a disability claim or receiving workman's compensation or seeking either as a result of their low back pain;
* Diagnosis of current depression or psychiatric disorder requiring treatment, or such a diagnosis in the previous 6 months;
* Beck Depression Inventory (BDI) Ia score greater or equal to 19 for two consecutive completions; if the first score meets this criteria, the participant must be re-tested before his/her next visit, but if the second score does not meet this criteria, the participant will be included and followed closely throughout the study
* Use of therapeutic doses of antidepressant medications (i.e., tricyclic depressants, SSRIs, SNRIs; low doses used for sleep may be allowed);
* Significant other medical disease such as unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy;
* History of gastrointestinal ulcer during the past year;
* History of myocardial infarction in the past year;
* Uncontrolled hypertension;
* Renal insufficiency;
* Allergic to, or non-tolerant of, NSAIDs;
* History of aspirin-sensitive asthma;
* Current use of recreational drugs or history of alcohol or drug abuse;
* Any change in medication for back pain in the last 30 days only applicable for visit 1
* High dose opioid prophylaxis, as defined as > 50mg morphine equivalent/day;
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
* Evidence of poor treatment compliance, in the judgment of the investigator;
* Intra-axial implants (e.g. spinal cord stimulators or pumps);
* All exclusion criteria for MR safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia;
* Pregnancy, or inability to use an effective form of contraception in women of child-bearing age;
* Diabetes (Type I or Type II);
* Lactose intolerance or sensitivity to lactose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apkar V Apkarian, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vachon-Presseau E, Abdullah TB, Berger SE, Huang L, Griffith JW, Schnitzer TJ, Apkarian AV. Validating a biosignature-predicting placebo pill response in chronic pain in the settings of a randomized controlled trial. Pain. 2022 May 1;163(5):910-922. doi: 10.1097/j.pain.0000000000002450. PMID 34433773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Treatment Intervention | Active Treatment Intervention | Placebo Treatment Intervention
Started | 14 | 40 | 40
Completed | 11 | 33 | 33
Not Completed | 3 | 7 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1
Not completed — non compliance in phone ratings | 2 | 1 | 2
Not completed — undisclosed comorbidities | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment Intervention | Active Treatment Intervention | Placebo Treatment Intervention | Total
Number analyzed (Participants) | 14 | 40 | 40 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 31 | 33 | 75
  >=65 years | 3 | 9 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.6) | 58.0 (10.5) | 53.0 (14.3) | 55.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 23 | 17 | 49
  Male | 5 | 17 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 23 | 25 | 56
  White | 4 | 16 | 9 | 29
  More than one race | 2 | 0 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 40 | 40 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Pain Assessed by Visual Analogue Scale (VAS)
Description: Self-report pain using a VAS scale (0-10) : 0 represents no pain and 10 the worst imaginable pain.
  Results are presented as percentage (%) change in pain before and after the intervention (baseline and post-intervention, 12 weeks).
  Percentage change is calculated with post-intervention pain minus baseline pain, divided by baseline pain i.e. (post - baseline) / baseline.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage of pain change
Arm/Group | No Treatment Intervention | Active Treatment Intervention | Placebo Treatment Intervention
Number analyzed (Participants) | 11 | 33 | 33
percentage of pain change | -0.0145 (0.036) | -0.2082 (0.048) | -0.1109 (0.050)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: collected at each one of the 6 visits
Arm/Group | No Treatment Intervention | Active Treatment Intervention | Placebo Treatment Intervention
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 9/14 | 16/40 | 20/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Treatment Intervention (N=14) | Active Treatment Intervention (N=40) | Placebo Treatment Intervention (N=40)
pre-diabetic (Metabolism and nutrition disorders) | 1 | 0 | 0
Tooth Pain (General disorders) | 0 | 1 | 0
GI issues (Gastrointestinal disorders) | 0 | 1 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Seasonal allergies (General disorders) | 1 | 1 | 0
pain following injection (General disorders) | 1 | 0 | 1
human papillomavirus (Reproductive system and breast disorders) | 0 | 0 | 1
Sore throat (General disorders) | 0 | 0 | 1
Cortisone Shot in Right Hip (General disorders) | 0 | 1 | 0
Cataracts (Eye disorders) | 0 | 1 | 0
Cough (General disorders) | 1 | 0 | 2
Cold (General disorders) | 1 | 1 | 4
Cervical Cancer screening (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flu (Gastrointestinal disorders) | 0 | 1 | 1
High blood pressure (General disorders) | 0 | 2 | 0
Puncture Bruising (General disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Kidney Stones (Renal and urinary disorders) | 0 | 0 | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute pain in left latissimus dorsi (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Body Aches (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Acute infection (Infections and infestations) | 0 | 0 | 1
Molar tooth extraction (General disorders) | 0 | 0 | 1
Headache (General disorders) | 0 | 2 | 1
upset stomach (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Appetite Loss (General disorders) | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1
Cyst removal in left arm (General disorders) | 0 | 0 | 1
Right Latissimi dorsi Pain (General disorders) | 0 | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 2
Cystourethroscopy Procedure (Gastrointestinal disorders) | 1 | 0 | 0
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study has several limitations including:

1. The biosignature was poor predictability of individual participants' magnitude of pain relief, e
2. The univariate analyses suggest that some features of the model could be further optimized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT02986334/Prot_SAP_ICF_000.pdf